CLINICAL TRIAL: NCT02876757
Title: 5 Alpha Reductase Inhibitors And The Risk Of Suicide And Depression
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Other Study IDs: 2016 0906 192 000
Record Dates: First submitted 2016-08-05; First posted 2016-08-24 (Estimated); Results first posted 2018-02-05 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: BPH; Depression; Suicide
MeSH Terms: conditions — Depression; Suicide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 5ARI Users
  Interventions: Drug: 5ARI
- Non 5ARI users

INTERVENTIONS:
Drug: 5ARI — Exposure to finasteride/dutasteride
  Groups: 5ARI Users

SUMMARY:
In December 2015, Health Canada issued a warning about a potential relationship between suicide and finasteride use and called for further research. No population based studies have assessed the risk of suicide with finasteride use, and this risk is not currently part of the product monograph. Furthermore, the link between depression and finasteride has not been well studied in the older population who are the primary users of this medication.

ELIGIBILITY:
Inclusion Criteria:

* All men >66 years of age in Ontario between 2003-2013

Exclusion Criteria:

* Non Ontario residents
* No prescriptions filled in prior 180 days
* Prior exposure to finasteride/dutasteride in the 2 years prior to study enrollment.
* Prescription initiated during hospital admission or ER visit.

Ages: 66 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All men >66 years of age in Ontario between 2003-2013
Sampling Method: Non-Probability Sample
Enrollment: 186394 (Actual)
Dates: Start 2003-01; Primary Completion 2013-12 (Actual); Study Completion 2017-03 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 5ARI Users | Non 5ARI Users
Started | 93197 | 93197
Completed | 93197 | 93197
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Non 5ARI Users: Matched patients without 5ARI usage
- Total: Total of all reporting groups
Arm/Group | 5ARI Users | Non 5ARI Users | Total
Number analyzed (Participants) | 93197 | 93197 | 186394
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.6 (6.7) | 75.5 (6.9) | 75.5 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 93197 | 93197 | 186394
Region of Enrollment [Number; unit: participants]
  Canada | 93197 | 93197 | 186394
Prior depression [Count of Participants; unit: Participants] | 3353 | 3353 | 6706

OUTCOME MEASURES:

1. Primary Outcome: Suicide (Based on Administrative Data Elements From Ontario Registrar General Death Database, National Ambulatory Care Reporting System, Hospital Discharge Abstracts, and Ontario Regional Mental Health Database)
Description: 1. Ontario Registrar General Death database. Use the COD_primary variable (used from 2003 onwards) to define suicide, based on an ICD10 code of X60-X84.
  2. NACRS: X60-84 (dx10code1-dx10code10) AND dead on arrival or death after arrival (visdisp2002 = 10 or 11). Consider admission date the date of the event.
  3. OMHRS: Discharge reason (dischreason (X90) = 2). Died from suicide. Consider admission date the date of the event.
  4. CIHI-DAD (Consider admission date the date of the event):
  i. suicide=1, or ii. dx10code1-25= ICD10 X60-84 AND dischdisp="07".
Time Frame: Through study completition, an average of 18 months.
Measure: Count of Participants; unit: Participants
Arm/Group | 5ARI Users | Non 5ARI Users
Number analyzed (Participants) | 93197 | 93197
Participants | 38 | 36

2. Secondary Outcome: Suicide Attempt (Based on Administrative Data Elements From National Ambulatory Care Reporting System, and Ontario Regional Mental Health Database)
Description: 1. NACRS: presentation to the emergency room: ICD 10 codes X60-X84 (intentional self harm).
  2. OMHRS: admission with suicide ideation.
  i. Self injury attempts: D1A or selfinjury_attempt=3, 4, 5, or 6 ii. Self injury intent: D1B or selfinjury_intent=1 iii. Self injury considered: D1C or selfinjury_cons=3, 4, 5 or 6 iv. Self injury plan: D1DB or suicide_plan=1
Time Frame: Through study completition, an average of 18 months.
Measure: Count of Participants; unit: Participants
Arm/Group | 5ARI Users | Non 5ARI Users
Number analyzed (Participants) | 93197 | 93197
Participants | 169 | 130

3. Secondary Outcome: Depression (Based on Administrative Data Elements From Hospital Discharge Abstract Database, and Ontario Regional Mental Health Database and Ontario Health Insurance Plan)
Description: 1. Any CIHI-DAD/SDS ICD 10 code, OR
  2. Any OMRHS code Axis1_dsm4code1-19 or Axis2_dsm4code 1-7 OR
  3. Look for any OHIP record billed by Mainspecialty = "PSYCHIATRY" with a diagnosis of depression OHIP dxcode 311, OR
  4. ≥2 GP visits within 2 years AND both with OHIP dxcode 311
  i. OHIP dxcode: 311 ii. ICD 10: F32.0, F32.1, F32.2, F32.3, F32.8, F32.9, F33.0, F33.1, F33.2, F33.3, F33.4, F33.8, F34.1 iii. Psychiatry visits defined as any of these OHIP fee codes: A195, A895, A190, A795, A695, A395, A196, A193, A194, A191, A192 iv. OMHRS: 29620-29626, 29630-29636, 31100 (major depressive disorder)
Time Frame: Through study completition, an average of 18 months.
Population: This population is restricted to those who had no history of depression, thus it is a subgroup of the total study population.
Measure: Count of Participants; unit: Participants
Arm/Group | 5ARI Users | Non 5ARI Users
Number analyzed (Participants) | 89844 | 89844
Participants | 1750 | 1231

ADVERSE EVENTS:
Description: Please note that only mortality from suicide was assessed, all-cause mortality could not be determined.
Groups:
- Non 5ARI Users: Matched control patients with no exposure to 5ARI
Arm/Group | 5ARI Users | Non 5ARI Users
All-Cause Mortality (participants affected / at risk) | 160/93197 | 139/93197
Serious Adverse Events (participants affected / at risk) | 0/93197 | 0/93197
Other Adverse Events (participants affected / at risk) | 0/93197 | 0/93197

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No